CLINICAL TRIAL: NCT05575336
Title: Integrated Personalized Care for Patients with Advanced Chronic Diseases to Improve Health and Quality of Life
Brief Title: Assessment of the Effectiveness, Socio-economic Impact and Implementation of a Digital Solution for Severe Patients
Acronym: ADLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosistemak Institute for Health Systems Research (Other)
Collaborators: NHS Lanarkshire (Other Government); Odense University Hospital (Other); Assuta Ashdod Hospital (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Gesunder Werra-Meißner-Kreis GmbH (Unknown); Maccabi Healthcare Services, Israel (Other); Osakidetza (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 875209
Record Dates: First submitted 2022-09-22; First posted 2022-10-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV; Chronic Obstructive Pulmonary Disease Severe
Keywords: Advanced chronic conditions; NYHA III-IV; >2 GOLD Scale; Multimorbidity; Personalized care; Integrated care; Early detection; Clinical decision support services; Patient and informal caregiver empowerment; Shared decision making; Patient Reported Outcome Measures (PROMs); Outcome-based care; Quality of life

STUDY DESIGN:
Intervention Model Description: A quasi-experimental trial following a multicentre, non-randomized, non-concurrent, unblinded and controlled design. Patients belonging to the intervention group will be under the ADLIFE intervention, while patients on the control group will follow the standard of care (SoC). The mixed-method approach will provide scientific evidence based on the effectiveness, socio-economic, implementation and technology acceptance assessment of ADLIFE intervention compared to the SoC when applied in real-life settings. The quantitative outcomes will be analysed not only at the individual level but also at the health organisation level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Use of the ADLIFE system
  Interventions: Other: ADLIFE intervention
- Control group (No Intervention): Patients will receive the Standard of Care

INTERVENTIONS:
Other: ADLIFE intervention — The ADLIFE toolbox will be deployed, used and evaluated in seven healthcare environments to demonstrate the effectiveness of the ADLIFE intervention in clinical real conditions. Patients participating in ADLIFE will have a personalised care plan, created in the ADLIFE toolbox, developed and managed together with their healthcare professionals. PCPMP will be used within clinical sites´ ICT systems to create patient care plans based on most recent clinical data, following clinical evidence. The main task of patients and informal caregivers will be to use the ADLIFE toolbox as part of their healthcare process together with their healthcare professionals.
  Patients recruited will use the ADLIFE system during the pilot study for a follow-up period between 3 and 12 months.
  Arms: Intervention group

SUMMARY:
ADLIFE is a EU-funded project developing innovative digital health solutions to support healthcare planning and care delivery for patients with advanced chronic conditions (chronic obstructive pulmonary disease and/or heart disease failure). ADLIFE's technology innovations will be deployed, used and evaluated in seven healthcare environments in Spain, the UK, Sweden, Germany, Denmark, and Israel.

ADLIFE intends to impact three stakeholders: patients, informal caregivers and health professionals, and consequently across the seven participating international healthcare systems. ADLIFE intervention aims at slowing down the patients' functional deterioration, ensuring their quality of life and promoting shared decision making, reducing the caregiver burden, and improving the health professional working conditions; all this under the scenario of an improvement in the healthcare resource use.

The research aims to prove whether the ADLIFE intervention can deliver appropriate targeted and timely care for patients with severe long-term diseases when applied in real-life settings. Based on a mixed-method approach, the study will provide scientific evidence based on the effectiveness, socio-economic, implementation and technology acceptance assessment of ADLIFE compared to the standard of care (SoC) to provide scientific evidence supporting the funding decision-making of the ADLIFE intervention.

DETAILED DESCRIPTION:
The ADLIFE project (GA 875209) is funded by the EC and Co-ordinated by Kronikgune Institute for Health Services Research. The consortium is made up of a total of 12 partners, supplying technical, clinical & research expertise. These partners are based in the UK, Spain, Sweden, Denmark, Turkey, Israel, Poland, Belgium and Germany.

The research project ADLIFE aims to develop and implement innovative, personalised and digital solutions for the integrated healthcare of elderly people with advanced chronic diseases, especially for patients with COPD and/or chronic heart failure (www.adlifeproject.com). The digital solutions (ADLIFE toolbox) involves two interconnected platforms: the Patient Empowerment Platform (PEP), used by patients and informal caregivers and the Personalised Care Plan Management Platform (PCPMP) used by healthcare professionals. In addition, PCPMP includes a Service to assist clinical decision support (CDSS).

The work plan of the project is structured in three phases. The 1st phase addresses the Organizational issues and ICT platforms implementation. The 2nd phase focuses on the Intervention's large-scale deployment. ADLIFE intervention will be implemented in seven regions representing six different countries, involving patients, informal caregivers and healthcare professionals. The 3rd and last phase will conduct an evaluation where ADLIFE scientific question will be answered. The main research question is - "When applied in real-life settings, is the use of the ADLIFE toolbox able to deliver appropriate targeted and timely care for patients with Advanced Chronic Diseases?". Care will be considered appropriate when it is deployed at the time and in the way is needed in order to generate the best possible gain in health and quality of life. The scientific question reflects the complex innovation intervention and three complementary evaluation approaches will be used:

* An effectiveness assessment will be conducted to estimate the ADLIFE intervention impact compared to the Standard of care, applying mixed methods combining quantitative and qualitative analysis.
* A socio-economic impact assessment will estimate the long-term economic impact of the ADLIFE intervention compared to the Standard of care, applying a budget impact analysis based on simulation modelling.
* An implementation assessment will be performed under three different perspectives: the implementation of the research project itself will be assessed as well as the contextual factors that are relevant for the translation of the innovation action into routine practice and the acceptance of the technology and adoption evaluation.

The study is aiming to recruit a minimum of 846 patients, 1183 informal caregivers and 679 healthcare professionals to the ADLIFE pilot study across all seven pilot sites. in Basque Country (Osakidetza), United Kingdom (National Health Service Lanarkshire and University Hospital Coventry & Warwickshire - National Health Service Trust), Denmark (Odense University Hospital), Germany (Gesunder Werra-Meißner Kreis), Sweden (Region Jämtland Härjedalen) and Israel (Assuta Ashdod Hospital - Maccabi Healthcare Services Southern Region).

The ADLIFE intervention consists of the deployment and use of the ADLIFE toolbox by patients, informal caregivers and health professionals in the aforementioned pilot settings. The intervention starts in December 2022. The project envisages a three-month window from the start of the intervention to achieve the total number of patients recruited. During the study period, patients will have a personalised care plan, created in the ADLIFE toolbox, which will be developed and managed together with their healthcare professionals. The main task of patients and informal caregivers will be to use the ADLIFE toolbox as part of their healthcare process together with their healthcare professionals. All participants will be trained in the use of the platforms and their participation prior to the start of the study. The intervention will end in November 2023, after which the evaluation will be carried out to analyse the feasibility and benefits of the ADLIFE solution.

ADLIFE will comply with the data protection legislation of the European Union GDPR and additional legislation in each country on health care data and medical research. Informed consent to participate in the study will be obtained from intervention patients. The patients who are recruited will receive care and treatment using the ADLIFE system, will have identifiable data collected about them by healthcare professionals in PCPMP, and will use, and provide information about themselves, in the PEP system. In addition to the clinical data captured, the intervention group patients, their carers and the healthcare professionals involved in the project will participate in a series of system/project evaluations before and after the study.

A separate cohort of patients will be identified retrospectively from local health records at the end of the study to create a 'control' group. These patients will match the same inclusion criteria. However, this control group will have no active role in the study (they will follow the standard of care of their organization) and only their anonymised data will be utilized so that health-related outcomes, resource utilisation, medication use, etc., can be compared for the two groups over the same period.

Evaluation analyses will be carried out with control data and intervention data collected in each pilot site. The data for project evaluation purposes will only be available to the site from which the data originated, it will be kept within the healthcare provider infrastructure. For the evaluation process, these data will be coded protected in order to reduce risks. The healthcare utilisation and outcome data collected from intervention patients will be extracted from the ADLIFE system itself in a pseudonymised format. Data from control data will be collected from local health records systems in an anonymized format. The relevant individual-level data for study evaluation will be processed and will be sent to the evaluation partners to carry out the clinical evaluations of the ADLIFE solution.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS-Inclusion criteria

* Senior (over 55)
* Heart failure (NYHA III-IV) in functional stage III/IV according to the NYHA scale and stages C and D of the ACCF/AHA classification. Stable phase (at least two months without decompensation requiring hospital care)
* And/or COPD (FEV1<50), >2 GOLD scale, and/or mMRC ≥ 2 and/or CAT ≥ 10 and/or use of oxygen at home
* With or without comorbidities
* They are able to provide informed consent
* They still live and generally plan on living in their home for the intervention duration
* They or their informal caregivers are able to use digital technology, communication tools, and/or networks and have access to a computer, laptop, tablet or smartphone and wifi/internet connection.
* They or their informal caregivers understand, read and talk the native language.

INFORMAL CAREGIVERS- Inclusion criteria

The informal caregiver will be a person who provides occasional or regular support to the patient's needs. Caregivers are eligible if:

* The patients they care for meet the inclusion criteria
* They give consent to participate

HEALTHCARE PROFESSIONALS-Inclusion criteria

Healthcare professionals are eligible if they care for patients who meet the inclusion criteria and consent to participate. Healthcare professionals taking part in ADLIFE should be:

* involved in the selected patients' care.
* open to new ways of working, specifically as part of coordinative and collaborative teams.
* open to the use of new technology. They should be willing to learn how to use technology to support their work.

Exclusion Criteria:

PATIENTS-Exclusion criteria

Patients are not eligible for recruitment if:

* Presence of active malignant neoplastic disease.
* Inclusion in the active list of any kind of transplantation.
* No signature of Informed consent by a legally capable patient.
* Patients who have participated in ADLIFE and later have withdrawn from their participation in the study the intervention formally are not eligible for recruitment again.

INFORMAL CAREGIVERS-Exclusion criteria

-Caregivers are not eligible if the patients they care for meet the exclusion criteria.

HEALTHCARE PROFESSIONALS-Exclusion criteria

* Healthcare professionals are not eligible if they do not care for patients who meet the inclusion criteria or only care for patients who meet the exclusion criteria.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline patient visits to the emergency (ER) department at the follow-up period (3-12 months) | The primary outcome will be observed for the follow-up period, 3-12 months after the baseline.
  Change from Baseline in the number of patient visits to the emergency (ER) department during the follow-up month-period. Data collected from EHR.

SECONDARY OUTCOMES:
Change from baseline Patient-Reported Outcome Measurements (PROMs) on health-related quality of life at the follow-up period (3-12 months) | The change in the health related quality of life of the patient measured by means of EQ-5D-5L will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measure reported by patients by means of completion of the questionnaire EQ-5D-5L
Change from baseline PPatient-Reported Outcome Measurements (PROMs) on mood/emotional health at the follow-up period (3-12 months) | The change in the mood/emotional health of patient measured by means of HADS-Hospital Anxiety and Depression Scale will be observed for the follow-up period (3-12 months), starting from the baseline.
  Outcome measure reported by patients by means of completion of the questionnaire HADS-Hospital Anxiety and Depression Scale
Change from baseline Patient-Reported Outcome Measurements (PROMs) on the ability of patients to perform tasks that are required to live independently in the community measured by Lawton scale at the follow-up period (3-12 months) | The change on the ability of patients to perform tasks that are required to live independently in the community measured by means of Lawton scale will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measure reported by patients by means of completion of the Lawton scale
Change from baseline capability of the patient to perform basic activities in daily life at the follow-up period (3-12 months) | The change on the capability of the patient to perform basic activities in daily reflecting the ability to function independently life measured by means of Barthel index will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measured reported by patients by means of answering of the Barthel Index
Change from baseline Patient-Reported Outcome Measurements (PROMs) on health status in patients with heart failure at the follow-up period (3-12 months) | The change on health status in patients measured by means Kansas City Cardiomyopathy Questionnaire score questionnaire will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measure reported by patients by means of completion of the questionnaire Kansas City Cardiomyopathy Questionnaire score
Change from baseline Patient-Reported Outcome Measurements (PROMs) on the impact of COPD on the patients' health status at the follow-up period (3-12 months) | The change on the impact of COPD on the patient's health status measured by means of COPD assessment test score will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measure reported by patients by means of completion of the questionnaire COPD assessment test score
Change from baseline Patient-Reported Outcome Measurements (PROMs) on complexity at the follow-up period (3-12 months).. | The change on the complexity measured by means of Modified Medical Research Council -mMRC- Dyspnea Scale will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measure reported by patients by means of completion of the Modified Medical Research Council -mMRC- Dyspnea Scale
Resource use due to patient healthcare visits | Resource use of intervention patients will be measured during the 12-months before the baseline and during the follow-up period (3-12 months)
  Outcome measured by means of number and type of patient healthcare visits
Resource use due to number of patient hospital admissions | Resource use of intervention patients will be measured during the 12-months before the baseline and during the follow-up period (3-12 months)
  Outcome measured by means of the number of patient hospital admissions
Resource use due to duration of patient hospital admissions | Resource use of intervention patients will be measured during the 12-months before and after the baseline
  Outcome measured by means of the number of the days of the patient hospital admissions
Associated costs to resource use due to number and type of patient healthcare visits | Resource use of intervention patients will be measured during the 12-months before the baseline and during the follow-up period (3-12 months)
  Outcome measured by cost of patient healthcare visits (considering the number, duration and the unit costs)
Associated costs to resource use due to patient hospital admissions | Resource use of intervention patients will be measured during the 12-months before the baseline and during the follow-up period (3-12 months)
  Outcome measured by cost of patient hospital admissions (taking into account the number, duration and the unit costs of hospitalisations)
Change from baseline burden of care of the informal caregivers at the follow-up period (3-12 months) | The change on the Burden of care measured by means of Zarit Burden Interview will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measured by completion of Zarit Burden Interview, ZBI by the informal caregivers
Associated costs to drug prescription | Resource use of intervention patients will be measured during the 12-months before the baseline and for the follow-up period (3-12 months)
  Outcome measured by total drug prescription cost that patients have
Change from baseline Technology acceptance and future adoption of the ADLIFE intervention by ADLIFE participants (patients, informal caregivers and health care professionals) after the follow-up period | The change on the technology acceptance measured by means of the Unified Theory of Acceptance and Use of Technology will be observed for the follow-up period (3-12 months), starting from the baseline
  Outcome measured by completion of the Unified Theory of Acceptance and Use of Technology (UTAUT)
Satisfaction with accessibility, security and Personalized Care Plans by ADLIFE participants (patients, informal caregivers and health care professionals) | The satisfaction with accessibility, security and Personalized Care Plans measured by means of semi-structured interviews will be observed after follow-up period (3-12 months) from the baseline
  Outcome measured by qualitative analyses (semi-structured interviews)
Barriers/facilitators related to the implementation process, by ADLIFE participants (patients, informal caregivers and health care professionals) | The change on the barriers/facilitators related to the implementation process measured by means of semi-structured interviews will be observed after the follow-up period (3-12 months) from the baseline
  Outcome measured by qualitative analyses (semi-structured interviews)
Perceived coordination among settings by health care professionals | The change on the perceived coordination among settings measured by means of semi-structured interviews will be observed after the follow-up period (3-12 months), from the baseline
  Outcome measured by qualitative analyses (semi-structured interviews)
Quality of care related to integration of care, decision making process and working condition by health care professionals | The change on the quality of care related to integration of care, decision making process and working condition measured by means of semi-structured interviews will be observed after the follow-up period (3-12 months), from the baseline
  Outcome measured by qualitative analyses (semi-structured interviews)
Perceptions on healthcare visits and hospital admissions burden by health care professionals | The change on the perceptions on healthcare visits and hospital admissions burden measured by means of semi-structured interviews will be observed after 12 months from the baseline
  Outcome measured by qualitative analyses (semi-structured interviews)
Implementation assessment by health care professionals, IT staff and clinical managers | The change on the implementation assessment measured by means of semi-structured interviews will be observed after 12 months from the baseline.
  Outcome measured by contextual factors focusing on local technological, organizational, and human factor (semi-structured interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban de Manuel, Study Chair — Instituto de Investigación en Servicios de Salud KRONIKGUNE
Locations (7):
- Odense University Hospital, Odense, Region Syddanmark, Denmark
- Gesunder Werra-Meißner-Kreis GmbH, Eschwege, Hesse, Germany
- Israel (2):
  - Maccabi Healthcare Services Southern Region, Ashdod
  - Assuta Ashdod Hospital, Ashdod
- Osakidetza, Vitoria-Gasteiz, Araba, Spain
- United Kingdom (2):
  - UNIVERSITY HOSPITALS COVENTRY AND WARWICKSHIRE NHS Trust, Coventry, Warwickshire
  - NHS Lanarkshire, Glasgow

IPD SHARING:
Plan to Share IPD: No